CLINICAL TRIAL: NCT01909895
Title: Translational Research of Negative Emotions and Acute Endothelial Dysfunction
Brief Title: Study of the Effects of Negative Emotions on Endothelial Function
Acronym: PUME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daichi Shimbo, Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AAAK4250; 1R01HL116470-01 (NIH)
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Emotions; Endothelial Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anger induction (Experimental): The participant will be asked to undergo a validated anger induction task.
  Interventions: Other: Anger Induction
- Depressed Mood Induction (Experimental): The participant will be asked to undergo a validated depression/sadness induction task.
  Interventions: Other: Depressed Mood Induction
- Anxiety Induction (Experimental): The participant will be asked to undergo a validated anxiety induction task.
  Interventions: Other: Anxiety Induction
- Neutral emotion task (Other): The participant will be asked to undergo a validated neutral task (i.e. count aloud by ones, starting with one and ending with 100, over and over, until the task period has ended).
  Interventions: Other: Neutral emotion task

INTERVENTIONS:
Other: Anger Induction — The participant is asked to recall an incident in the recent past during which they became moderately to extremely angry, or is asked to read statements out loud evoking moderate to extreme feelings of anger. The participant is asked to take a few moments to bring the details of the incident to mind and, when ready, to describe the incident in great detail to the experimenter. Participants are asked to describe key elements, such as any dialogue that transpired during the incident, along with other details of the incident, particularly regarding the feelings of that particular emotion experienced at the time. In so doing, the experimenter works to re-elicit the emotions that accompanied the original incident. The duration of the negative emotion induction task is 8 minutes.
  Arms: Anger induction
Other: Depressed Mood Induction — The participant will be asked to undergo a validated depression/sadness induction task.
  Arms: Depressed Mood Induction
Other: Anxiety Induction — The participant will be asked to undergo a validated anxiety induction task.
  Arms: Anxiety Induction
Other: Neutral emotion task — This is a neutral control task that each of the negation emotion induction tasks will be compared to.
  Arms: Neutral emotion task

SUMMARY:
Study aims and hypotheses are as follows:

Primary Hypotheses:

Compared to the neutral condition, the anger recall task will acutely induce endothelial dysfunction by impairing endothelium-dependent arterial vasodilation (Hypothesis 1a); increasing circulating levels of EC-derived microparticles (EMPs), a marker of EC injury (Hypothesis 1b); and reducing circulating levels of bone marrow-derived endothelial progenitor cells (EPCs), a marker of EC reparative capacity (Hypothesis 1c).

Secondary Hypotheses:

Compared to the neutral condition, the depressed mood and separately the anxiety recall tasks will acutely impair endothelium-dependent arterial vasodilation, increase circulating levels of EMPs, and reduce circulating levels of bone marrow-derived EPCs. There will be a relation of the level of self-reported anger, depressed mood, and anxiety with endothelial dysfunction.

DETAILED DESCRIPTION:
Atherosclerosis-related cardiovascular disease (CVD) events remain the leading causes of morbidity and mortality in industrialized nations. Atherosclerosis is a diffuse disease characterized by the deposition of lipid and other blood-borne material within the arterial wall. Evidence demonstrates that disruption of an arterial atherosclerotic plaque and subsequent thrombus formation is responsible for the onset of CVD events. Cardiovascular research efforts have been directed toward the identification of early underlying factors that initiate this cascade.

It has been known for some time that the experience of negative emotions is associated with an increased risk of incident CVD events, independent of traditional risk factors. Among the best-studied negative emotions is anger. Population-based studies have demonstrated that the experience of anger is a trigger of incident CVD events. The mechanism(s) by which provoked anger acutely affects the pathways that underlie atherosclerosis development and progression remain to be fully characterized.

Endothelial dysfunction is a promising mechanism that may explain the link between anger and incident CVD events. Vascular endothelial cells (ECs) play essential roles in maintaining vascular tone and the integrity of blood vessels. Evidence suggests that endothelial dysfunction is an early pathogenic process underlying atherosclerosis development and CVD event onset. Our preliminary findings show in apparently healthy individuals, an anger recall task acutely induces endothelial dysfunction by impairing endothelium-dependent vasodilation, injuring ECs, and disrupting the molecular processes underlying EC reparative capacity. We have additionally found that this task may induce endogenous nitric oxide (NO) inhibition, which plays a central role in aggravating endothelial dysfunction. Therefore, NO inhibition may partially mediate anger-provoked endothelial dysfunction.

Although the strongest data are on anger-provoked CVD events, there is also some evidence that the experience of other core negative emotions such as depressed mood and anxiety may trigger CVD events. Whether the provocation of depressed mood and anxiety acutely induces endothelial dysfunction and NO inhibition remains to be determined. The overall aim of this study is to primarily examine the acute effects of provoked anger and secondarily depressed mood and anxiety on EC health. We will also explore whether NO inhibition partially mediates the acute effects of anger, depressed mood, and anxiety on endothelial function. Examination of these critical pathways will help identify the biological pathways by which the experience of core negative emotions leads to incident CVD risk.

To address these highly significant research questions, we propose a state-of-the-art, laboratory-based, randomized controlled experiment in which 280 participants will be randomized to one of four experimental conditions: an anger recall task (N=70), a depressed mood recall task (N=70), an anxiety recall task (N=70), and an emotionally neutral condition (N=70).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Fluent in English

Exclusion Criteria:

* History of any chronic medical condition including prevalent CVD and traditional risk factors
* Active smoking
* Chronic medication use, including over-the-counter drugs or herbal medications
* History of psychosis, a mood disorder, or any overt personality disorder
* Latex allergy
* Poor peripheral veins with low possibility of getting IV access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent arterial vasodilation | baseline
Circulating EMPs expressing CD62E | baseline
Circulating early EPCs (KDR+, CD34+, CD133+ cells) | baseline
Endothelium-dependent arterial vasodilation | 3 mins after end of mood induction
Endothelium-dependent arterial vasodilation | 40 mins after end of mood induction
Endothelium-dependent arterial vasodilation | 70 mins after end of mood induction
Endothelium-dependent arterial vasodilation | 100 mins after end of mood induction
Circulating EMPs expressing CD62E | 3 mins after end of mood induction
Circulating EMPs expressing CD62E | 40 mins after end of mood induction
Circulating EMPs expressing CD62E | 70 mins after end of mood induction
Circulating EMPs expressing CD62E | 100 mins after end of mood induction
Circulating early EPCs (KDR+, CD34+, CD133+ cells) | 3 mins after end of mood induction
Circulating early EPCs (KDR+, CD34+, CD133+ cells) | 40 mins after end of mood induction
Circulating early EPCs (KDR+, CD34+, CD133+ cells) | 70 mins after end of mood induction
Circulating early EPCs (KDR+, CD34+, CD133+ cells) | 100 mins after end of mood induction

SECONDARY OUTCOMES:
Circulating EMPs expressing CD31 | baseline; 3 mins, 40 mins, 70 mins, 100 mins after end of mood induction
Circulating EMPs expressing CD51 | baseline; 3 mins, 40 mins, 70 mins, 100 mins after end of mood induction
Self-reported anger, depressed mood, and anxiety | baseline; 3 mins, 40 mins, 70 mins, 100 mins after end of mood induction

OTHER OUTCOMES:
Nitric oxide(NO) inhibition | baseline; 3 mins, 40 mins, 70 mins, 100 mins after end of mood induction
  Circulating measures of asymmetric dimethylarginine (ADMA) and oxidative stress measures
Stress response | baseline; 3 mins, 40 mins, 70 mins, 100 mins after end of mood induction
  Circulating measures of catecholamines, cortisol, endothelin-1; blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Daichi Shimbo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ensari I, Burg MM, Diaz KM, Fu J, Duran AT, Suls JM, Sumner JA, Monane R, Julian JE, Zhao S, Chaplin WF, Shimbo D. Putative mechanisms Underlying Myocardial infarction onset and Emotions (PUME): a randomised controlled study protocol. BMJ Open. 2018 May 31;8(5):e020525. doi: 10.1136/bmjopen-2017-020525. PMID 29858417